CLINICAL TRIAL: NCT00444236
Title: Effect of Acid Reflux on Respiratory Physiology During Exercise in Athletes With GER-Response to Acid Suppression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study due to slow enrollment.
Sponsor: University of Utah (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Kathryn A. Peterson, MD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB # 20135; Exercise/Asthma
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Exercise Triggered Asthma; Gastroesophageal Reflux
Keywords: asthma; GERD; reflux; exercise
MeSH Terms: conditions — Gastroesophageal Reflux; Asthma; Motor Activity | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Nexium
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nexium — nexium or placebo 40 mg twice a day for 10-12 weeks. Therapy will then be switched for another 10-12 weeks
  Other Names: esomeprazole
  Arms: 1
Drug: Placebo — matching placebo for active drug
  Arms: 2

SUMMARY:
We propose that acid reflux affects respiratory dynamics (breathing) in patients who are exercising and that athletes improve their exercise capacity with acid suppression therapy. It is our intent to determine whether treatment of GER with strong acid suppression may alleviate symptoms, improve exercise capacity, and improve quality of life.

DETAILED DESCRIPTION:
This is a randomized, blinded, cross-over trial. We plan to take athletes with classical GER, cough, shortness of breath, chest tightness during exercise and subject them to complete pulmonary function testing in conjunction with exercise and pH testing. We will assess whether such athletes experience an increase in reflux duration and episodes during exercise. The athletes will be randomized (in a cross over fashion) to acid suppression (BID Nexium 40 mg) or placebo for 10-12 weeks. Both the athletes and investigators will be blinded. After 10-12 weeks, exercise testing (ramp protocol with VO2 and anaerobic threshold) with concurrent respiratory function testing will be repeated along with symptom assessment. After a brief washout period of 1-2 weeks, the athletes will then cross-over to the other study medication for 10-12 weeks. Again, at the end of the study period, symptomatic relief as well as respiratory function improvement will be assessed by repeating the initial exercise regimen. The exercise regimens during these medication regimens will not be held stable as indirectly, as a results of "feeling better or worse" from the medication/placebo, these patients may increase/ decrease their exercise routine, resulting in changes in their overall endurance, anaerobic threshold, etc (our endpoints). By keeping the regimen stable, we do not allow for the changes to occur which are large enough to detect.

ELIGIBILITY:
Inclusion Criteria:

* We plan to take athletes (cyclists) with GER (heartburn symptoms on a daily-weekly basis which are either improved by a trial of acid suppression or objectively documented via pH/endoscopic testing- this may include during exercise) who experience one or more of the following symptoms during exercise, limiting their perceived ability to exercise to full capacity:

  * choking
  * cough
  * wheezing
  * shortness of breath
  * chest tightness during exercise
* Athletes will be defined as persons who exercise on a routine basis (at least 3 times a week on average) for at least the past 6 months.
* Subjects must be at least 18 years old.

Exclusion Criteria:

* Pregnancy
* Age less than 18 years or greater than 65 years
* Abnormal methacholine challenge tests will not exclude one from enrollment as (has been documented in a prior study) often patients with GER will have heightened bronchial reactivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To assess whether acid suppression results in improvement in respiratory parameters in symptomatic patients. | 6 months

SECONDARY OUTCOMES:
To assess whether acid reflux events increase during exercise in athletes with symptomatic heartburn or respiratory discomfort during exertion. | 6 months
To assess whether long term acid suppression results in enhanced athletic performance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Peterson, MD, MSci, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States